CLINICAL TRIAL: NCT06200285
Title: International Hypothermia Registry: a Registry With Worldwide Cases of Accidental Hypothermia
Brief Title: International Registry of Accidental Hypothermia
Acronym: IHR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Evelien Cools, Medical Doctor, Principal Investigator, University Hospital, Geneva
Other Study IDs: 2022-02000
Record Dates: First submitted 2023-11-12; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Accidental Hypothermia
Keywords: Accidental Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood: Potassium, lactate, coagulation parameters, hemoglobin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Registry of patients with accidental hypothermia

SUMMARY:
Transient mild hypothermia (core body temperature 35-32°C) is common and usually without consequences for the brain or other organs. However, prolonged severe accidental hypothermia (core body temperature below 28°C) due to accidents is rare, and usually fatal in more than 50% of cases. Little is known on its physiopathology, on prognostic factors for rewarming decision or ideal rewarming techniques for better survival. Furthermore, complications after successful rewarming are extremely frequent and very often severe or fatal.

Accidental hypothermia is a frequent problem during the winter months and can be caused by snow sport accidents, near drowning and urban cold exposure. The International Hypothermia Registry's principle goal is to increase knowledge on accidental hypothermia by creating the largest database on accidental hypothermia which will comprise enough patient data to give a statistical power since the causes of accidental hypothermia and its treatment varies greatly.

The International Hypothermia Registry (IHR) will enable improvement of pre- and in-hospital treatment and rewarming methods, study survival predictors and prevention of post-rewarming complications. By this way, the IHR will permit the establishment of evidence-based diagnosis and treatment guidelines.

DETAILED DESCRIPTION:
The aim of the International Hypothermia Registry is to improve rescue, treatment and outcome of accidental hypothermia victims.

The principal objectives of the International Hypothermia Registry are:

* Improving the outcome of accidental hypothermic patients (survival and normal neurologic function);
* This outcome is dependent on the presenting status of the patient (temperature, trauma, cardiac arrest, etc.);
* The hospital treatment and rewarming method will also influence the outcome, invasive vs. non-invasive rewarming and rewarming rate.
* Quality control, assessment of hypothermia cases

This IHR is mainly prospective but retrospective entries are welcome.

There is no data limit on retrospective cases: cases of any year can be entered.

ELIGIBILITY:
Inclusion Criteria:

* Accidental hypothermia with body core temperatures equal or less than 35°C/95°F;
* Any cause leading to accidental hypothermia (e.g. mountain, water, urban);
* Any age, gender, or comorbidities;
* Any pre-hospital and hospital treatment and rewarming;
* Any outcome.

Exclusion Criteria:

* Patient opposition to be part of a study;
* Essential missing values, e.g. temperature.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators aim to include patients of any age.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-10-01 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2054-12 (Estimated)

PRIMARY OUTCOMES:
The Registry is a questionnaire, containing 252 variables divided into a demographical, prehospital, hospital and outcome section. The collected measurement data will be registered on REDCap. | through study completion, an average of 1 year
  For every patient, the questionnaire on REDCap will be filled in. Demographical data contain age, weight, consent status, ... . Prehospital data include the prehospital temperature, the circumstances of the accident (drowning, avalanche, intoxication, ... ), the presence of cardiac arrest, the first heart rhythm, ... . Hospital data contain the rewarming mode, the complications after and during rewarming. Outcome data cover the cerebral performance category after hospitalisation.
  Every further study with their specific outcomes using the data of the International Hypothermia Registry will be registered separately on clinical trials.gov. The data that are necessary to answer the scientific question defined in further studies will be extracted from REDCap.

CONTACTS AND LOCATIONS:
Locations (16):
- Austria (2):
  - Medical University Innsbruck, Innsbruck
  - Krankenhaus Barmherzige Brüder, Salzburg
- Rigshospitalet, Copenhagen, Denmark
- Klinik Immenstadt, Immenstadt im Allgäu, Germany
- Italy (3):
  - ASST Bergamo Est, Bergamo
  - EURAC Research, Bolzano
  - Ospedale Santa Chiara, Trento
- Hokkaido Ohno Memorial Hospital, Hokkaido, Japan
- Medical University of Silesia, Katowice, Poland
- Spain (2):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital de Cerdanya, Girona
- Switzerland (4):
  - Kantonsspital Chür, Chur
  - Division of Anaesthesiology, Geneva
  - Osepedale Regionale di Lugano, Lugano
  - University Hospital Zürich, Zurich
- University of Portsmouth, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://hypothermia-registry.org